CLINICAL TRIAL: NCT03094442
Title: Does Dexamethasone Administration Improve Recovery In Patients Undergoing Minimally Invasive Sacrocolpopexy?
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Eric Hurtado, Principal Investigator, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FLA 16-081
Record Dates: First submitted 2017-02-20; First posted 2017-03-29 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Quality of Life; Pelvic Organ Prolapse; Prolapses, Vaginal Vault
Keywords: Quality of Recovery; Minimally Invasive Sacrocolpopexy; Dexamethasone
MeSH Terms: conditions — Pelvic Organ Prolapse | interventions — Dexamethasone; Steroids; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dexamethasone (Active Comparator): Dexamethasone is a potent corticosteroid that has been widely used for chemotherapy induced nausea and vomiting. The mechanism of action is not completely understood. It has been proposed that a single dose may hinder the production and release of anti-inflammatory mediators. Dexamethasone also has a central antiemetic effect by inhibition of prostaglandin and/or release of endogenous opioids. A recent metanalysis concluded that Dexamethasone administration at induction is safe.
  We will be using a 8mg dose of Dexamethasone, that is equivalent to 2ml of injectable drug.
  Interventions: Drug: Dexamethasone
- Saline (Placebo Comparator): Normal saline contains 0.9% weight/ volume of sodium chloride. It is used routinely for intravenous resuscitation and fluid maintenance. Patients in the placebo arm will receive 2 ml of normal saline in the blinded syringe provided by the pharmacy.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Dexamethasone — An 8 mg dose of Dexamethasone is administered at the time of induction of general anesthesia. The medication is provided by the pharmacy in a blinded syringe.
  Other Names: Steroid
  Arms: Dexamethasone
Drug: Normal saline — Normal saline contains 0.9% weight/ volume of sodium chloride. It is used routinely for intravenous resuscitation and fluid maintenance. Patients in the placebo arm will receive 2 ml of normal saline in the blinded syringe provided by the pharmacy.
  Other Names: Placebo
  Arms: Saline

SUMMARY:
The primary aim is to evaluate whether standard administration of Dexamethasone at the time of general anesthesia induction at the time of minimally invasive sacrocolpopexy (MISC) would result in improved quality of recovery (QoR).

DETAILED DESCRIPTION:
There has been a public outcry regarding the continuing rise of health care expenditures. In 1997, the estimated costs of surgery for pelvic organ prolapse (POP) were $ 100.1 million. It is important to identify interventions that would improve the QoR in this patient population and to speed-up postoperative recovery. As most of these surgeries are performed in an outpatient manner as a 23 hour observation, improved recovery may also speed discharge and free-up valuable hospital resources.

Patients will receive either Dexamethasone or placebo ( normal saline) at the time of induction of general anesthesia. QoR questionnaires, Pain scale and postoperative nausea and vomiting scale (PONV).

ELIGIBILITY:
Inclusion Criteria:

1. Women over the age of 18
2. Women scheduled for minimally invasive sacrocolpopexy with or without concomitant anti-incontinence procedure and with or without concomitant hysterectomy
3. American Society of Anesthesiologists (ASA) class 1-2

Exclusion Criteria:

1. Daily use of steroids, antiemetics in the month prior to surgery
2. Chronic pain requiring daily opioid treatment
3. History of allergy/intolerance to Dexamethasone
4. ASA class 3
5. Numerical Pain score (NPS) of more than 4 at baseline
6. Renal/Liver disease
7. Diabetes mellitus
8. Pregnancy
9. Inability to answer questionnaires
10. Any systemic infections
11. Immuno compromised status

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Quality of recovery 40 (QoR-40) | baseline, 24 hours, 6 weeks
  Quality of Recovery 40 will be recorded at baseline, 24 hours and 6 weeks. The change in the mean scores will be computed for each group. The primary endpoint of change in QoR from baseline will be analyzed through t- test.

SECONDARY OUTCOMES:
Numerical Pain Scale | baseline, 24 hours, 6 weeks
  Pain at baseline, 24 hours and 6 weeks will be recorded.
Postoperative Nausea Vomiting Scale | 6 weeks
  Immediate nausea and vomiting 24 hours after surgery. Use of rescue antiemetics will be recorded

OTHER OUTCOMES:
postoperative urinary retention | 6 weeks
Infections | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: David Ossin, MD, Principal Investigator — Cleveland Clinic Florida
Locations (1):
- Cleveland Clinic Florida, Weston, Florida, United States

IPD SHARING:
Plan to Share IPD: No